CLINICAL TRIAL: NCT06385262
Title: Safety, Efficacy, and Tumor Immune Microenvironment Changes With Neoadjuvant Chemotherapy and Cemiplimab With or Without Alirocumab in Stage 1B-3A Non-Small Cell Lung Cancer: TOP 2301
Brief Title: TOP 2301: Neoadjuvant Chemo for NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Neal Ready MD PhD, Professor of Medicine, Duke University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00114645
Record Dates: First submitted 2024-04-22; First posted 2024-04-26 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — alirocumab; cemiplimab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Chemotherapy and cemiplimab (PD-1 inhibitor) every 3 weeks for 3 cycles with alirocumab (PCSK9 inhibitor) every 4 weeks prior to surgery
  Interventions: Drug: Alirocumab; Drug: Cemiplimab; Drug: Chemotherapy
- Arm B (Experimental): Chemotherapy and cemiplimab (PD-1 inhibitor) every 3 weeks for 3 cycles without alirocumab (PCSK9 inhibitor) prior to surgery
  Interventions: Drug: Cemiplimab; Drug: Chemotherapy

INTERVENTIONS:
Drug: Alirocumab — 300 mg subcutaneously every 4 weeks prior to surgery
  Arms: Arm A
Drug: Cemiplimab — 350mg IV every 3 weeks prior to surgery
Drug: Chemotherapy — Treating provider's choice of FDA approved platinum doublet chemotherapy IV every 3 weeks prior to surgery

SUMMARY:
In this open-label, two-arm, randomized phase 2 clinical trial, patients with clinical stage 1B-3A non-small cell lung cancer (NSCLC) will receive neoadjuvant chemotherapy and cemiplimab every 3 weeks for 3 cycles with or without alirocumab every 4 weeks prior to surgery.

Eligible patients will be randomized with equal allocation to two treatment groups. Permuted block randomization algorithm will be used for treatment assignment with stratification factors: stage (1B, 2A, 2B, 3A), and performance status (0 vs. 1).

The study hypothesis is that the addition of alirocumab to neoadjuvant chemoimmunotherapy will make tumor cells more immunogenic to cytotoxic T cells, resulting in an increase in complete pathologic responses in surgically resected tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Histological/cytological diagnosis of non-small cell lung cancer (NSCLC). Patient is eligible to enroll in the study based on clinical suspicion of NSCLC but are required to have a histological diagnosis of NSCLC in order to be eligible to receive treatment on study.
3. Clinical stage IB, IIA/IIB, or III (N0-2) amenable to surgical resection.
4. Primary tumor size of ≥ 3 cm (for all clinical stages to insure adequate tumor for correlative studies).
5. Agrees to research blood collections for study.
6. Deemed a surgical candidate.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. No prior chemotherapy, radiation therapy or biologic/targeted therapy for current diagnosis of lung cancer.
9. Measurable disease per Response Evaluation Criteria in Solid Tumours (RECIST) 1.1.
10. No active invasive malignancy in the past 2 years other than non-melanoma skin cancer. Cancers that are in-situ are not considered invasive.
11. Signed written informed consent including Health Insurance Portability and Accountability Act (HIPAA) according to institutional guidelines.
12. Sexually active males and females of reproductive potential must agree to use an appropriate contraceptive method during the study and for 120 days following the last dose of study drug.
13. Females of childbearing potential must test negative for pregnancy within 48 hours prior to any initial study procedure based on a serum pregnancy test. (If subject uses appropriate contraceptive methods from the time of the initial serum pregnancy test, then the subsequent pregnancy test can be done within 72 hours prior to start of study treatment. If appropriate contraceptive measures are not begun immediately with the first serum pregnancy test, then subsequent serum pregnancy tests must be done within 48 hours prior to the start of study treatment.)
14. Adequate organ function defined as:

    1. Absolute neutrophil count (ANC) ≥ 1500 per uL
    2. Platelets ≥ 100,000 per uL
    3. Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L without transfusion or growth factor dependency (within 7 days of assessment)
    4. Serum creatinine ≤ 1.5 x upper limit of normal (ULN) OR creatinine clearance (CrCl) or glomerular filtration rate (GFR) ≥ 60 mL/min for subject with creatinine levels > 1.5 x ULN
    5. Total bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
    6. Aspartate aminotransferase (AST) [serum glutamic-oxaloacetic transaminase (SGOT)] and alanine aminotransferase (ALT) [glutamic-pyruvic transaminase (SGPT)]≤ 2.5 x ULN
    7. Albumin ≥ 2.5 mg/dL
    8. International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy and within therapeutic range of intended use of anticoagulants
    9. Activated Partial Thromboplastin Time (aPTT) ≤1.5 x ULN unless subject is receiving anticoagulant therapy and within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

1. Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of study treatment.
2. Participants with known EGFR mutations, ALK translocation, or ROS1 translocation. If testing is done, an FDA-approved assay should be used.
3. Known history of active TB (Bacillus Tuberculosis).
4. Hypersensitivity to alirocumab or any of its excipients.
5. Concurrent administration of any other anti-tumor therapy.
6. Prior therapy with an anti-PD-1, anti-PD-L-1, or anti-PD-L2 agent.
7. Therapy with an anti-PCSK9 agent within 90 days of study entry.
8. Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
9. Inability to comply with protocol or study procedures.
10. Active infection requiring antibiotics, antifungal or antiviral agents, that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
11. Known history of, or any evidence of active, non-infectious pneumonitis.
12. Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or HCV infection; or diagnosis of immunodeficiency. Exceptions:

    1. Patients with HIV who have controlled infection (undetectable viral load and CD4 count above 350 either spontaneously or on a stable antiviral regimen) are permitted.
    2. Patients with HBV (hepatitis B surface antigen positive) who have controlled infection (serum hepatitis B virus DNA polymerase chain reaction (PCR) that is below the limit of detection AND receiving anti-viral therapy for hepatitis B) are permitted.
    3. Patients who are HCV antibody positive (HCV Ab +) who have controlled infection (undetectable HCV RNA by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) are permitted.
13. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency etc.) is not considered a form of systemic treatment. Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g. Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome and Myasthenia Gravis).
14. Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
15. Known additional invasive malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy in situ cervical cancer.
16. Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of study treatment.
17. Major surgery (other than definitive lung cancer surgery) within two weeks of study or other serious concomitant disorders that in the opinion of the investigator would compromise the safety of the patient or compromise the patient's ability to complete the study.
18. Any non-oncology, live vaccine therapy used for prevention of infectious diseases within 30 days prior to start of study treatment.

    Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines and are not allowed. Coronavirus Disease 2019 (COVID-19) vaccines are also allowed.
19. Myocardial infarction having occurred less than 6 months prior to study enrollment, any known uncontrolled arrhythmia, symptomatic angina pectoris, active ischemia, or cardiac failure not controlled by medications. Patients with coronary artery disease treated with surgery and/or stent > 6 months ago, if stable without symptomatic angina pectoris, active ischemia are eligible.
20. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
21. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either psychiatric or physical (e.g., infectious) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
Compare pathologic complete response (pCR) rate for neoadjuvant chemotherapy plus cemiplimab versus chemotherapy, cemiplimab, and alirocumab. | 2 years
  Pathologic complete response (pCR) is defined as a lack of all signs of cancer in tissue samples removed during surgery or biopsy after neoadjuvant therapy.

SECONDARY OUTCOMES:
Assess the preliminary efficacy of chemotherapy and cemiplimab with alirocumab as determined by objective response rate (ORR) | 2 years
  ORR is defined as complete response (CR) + major pathologic response (MPR) + partial response (PR)
Assess the preliminary efficacy of chemotherapy and cemiplimab with alirocumab as determined by disease-free survival (DFS) | 2 years
  Disease-free survival (DFS) is defined as the time from randomization to disease recurrence (first disease recurrence or death, whichever comes first) after surgery
Assess the preliminary efficacy of chemotherapy and cemiplimab with alirocumab as determined by overall survival (OS) | 2 years
  Overall survival (OS) is the length of time that a patient lives following treatment
Determine the safety of neoadjuvant chemotherapy and cemiplimab with alirocumab in early-stage non-small cell lung cancer (NSCLC) | 2 years
  Safety will be determined by evaluating the severe adverse events rate for the experimental therapy.
Determine the tolerability of neoadjuvant chemotherapy and cemiplimab with alirocumab in early-stage non-small cell lung cancer (NSCLC) | 2 years
  Tolerability will be determined by evaluating the severe adverse events rate for the experimental therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Ready, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No